CLINICAL TRIAL: NCT00514228
Title: Continuous Sunitinib Treatment in Patients With Unresectable Hepatocellular Carcinoma A Multicenter Phase II Trial
Brief Title: Sunitinib in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 77/06; SWS-SAKK-77/06; EU-20750; EUDRACT-2007-003977-22; CDR0000560441
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous sunitinib treatment (Experimental)
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — * Starting dose: 37.5 mg 3 x 12.5 mg capsule
  * Reduced dose: 25 mg 2 x 12.5 mg capsule
  Other Names: Sutent

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Demonstrate the antitumor activity of continuous sunitinib malate treatment in patients with unresectable hepatocellular carcinoma.

Secondary

* Evaluate the safety of sunitinib malate treatment.
* Measure serum cobalamin (i.e., vitamin B12) level during sunitinib malate treatment in order to investigate the relationship between sunitinib malate treatment and cobalamin deficiency.
* Control the cobalamin deficiency by cobalamin replacement.
* Investigate whether changes in tumor density could be used as a criterion for tumor response in future trials.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection on day 1 of each course to assess serum cobalamin levels and correlation with sunitinib malate treatment. Patients are also assessed for changes in tumor density and correlation with response. Baseline CT scans are compared with scans performed at 6 and 12 weeks to evaluate changes in CT-scan density due to tumor necrosis and response.

After completion of study therapy, patients are followed at least every 3 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically, cytologically, or radiologically confirmed hepatocellular carcinoma (HCC) meeting 1 of the following criteria:

  * Localized, surgically unresectable disease

    * Candidates for radical surgery for locally advanced disease are excluded
  * Metastatic disease
* Measurable disease, defined as ≥ 1 lesion, outside of pretreated areas, that can be measured in ≥ 1 dimension as ≥ 10 mm by spiral or multi-slice CT scan or MRI
* Child-Pugh class A or mildly decompensated Child-Pugh class B liver dysfunction

Exclusion criteria:

* Clinical ascites of any grade
* Clinical symptoms or history of CNS metastases or leptomeningeal disease
* Known fibrolamellar HCC or mixed cholangiocarcinoma and HCC

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-1
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* ALT ≤ 7 times ULN
* Albumin ≥ 2.5 g/dL
* Creatinine clearance ≥ 40 mL/min
* Quick test ≥ 50% (adequate coagulation)
* Urine dipstick for proteinuria < 2+ OR ≤ 1 g of protein in 24-hour urine collection
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy

Exclusion criteria:

* Pregnant or nursing
* Encephalopathy
* Malignancy within the past 5 years except for adequately treated cervical carcinoma in situ or localized nonmelanoma skin cancer
* Hemorrhagic or thrombotic cerebrovascular event in the past 12 months
* Documented variceal hemorrhage within the past 3 months
* History or presence of clinically significant acute or unstable cardiovascular, cerebrovascular, renal, gastrointestinal, pulmonary, immunological (except for the presence of hepatitis B virus, hepatitis C virus, or cirrhosis), endocrine, or central nervous system disorders
* Known HIV infection
* Active infection requiring IV antibiotics
* Arterial hypertension ≥ 150/100 mm Hg, despite therapy
* Ongoing cardiac dysrhythmias ≥ grade 2
* Atrial fibrillation of any grade
* Prolongation of QTc > 500 msec in screening ECG or history of familial long QT syndrome
* Inability to take oral medications
* Psychiatric disorder precluding understanding of information of study-related topics, giving informed consent, or interfering with compliance for oral drug intake

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* At least 4 weeks since prior surgery or liver-directed therapy (e.g., transarterial embolization/chemoembolization [limited to 5 treatments], radiofrequency ablation, cryoablation, radiotherapy, or percutaneous ethanol injection)

  * Previously treated lesions must remain separate from those to be measured in the present study
* Low-dose anticoagulants for maintenance of patency of central venous access or prevention of deep vein thrombosis allowed

Exclusion criteria:

* Prior systemic anticancer treatment for hepatocellular carcinoma
* Prior organ transplantation
* Treatment in a clinical study within the past 30 days
* Concurrent full-dose anticoagulant or requirement for anticoagulant therapy
* Concurrent experimental drugs or other anticancer therapy
* Concurrent use or anticipated need for CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, voriconazole, erythromycin, clarithromycin, and protease inhibitors)
* Concurrent CYP3A4 inducers (e.g., carbamazepine, continuous treatment with dexamethasone [> 2 mg/day for > 7 days], phenobarbital, phenytoin, rifampicin, and St John's wort)

  * Concurrent antacids allowed provided they are administered > 1 hour before or > 1 hour after study drug
* Concurrent elective major surgery
* Concurrent radiotherapy

  * Concurrent analgesic radiotherapy of nontarget lesions allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at 12 weeks

SECONDARY OUTCOMES:
Objective response | Objective response (CR+PR) to treatment will be determined. CR or PR is to be confirmed after a minimum of 4 weeks
Disease stabilization (DS) | Disease stabilization (CR, PR or SD) under sunitinib treatment will be determined
Duration of DS | Duration of DS (CR, PR or SD) will be calculated from the time that measurement criteria are met for the first time until documented tumor progression
Progression-free survival | PFS will be calculated from registration until documented tumor progression or death, whichever occurs first.
Time to progression | TTP will be calculated from registration until documented tumor progression or death due to tumor.
Overall survival | OS will be calculated from registration until death
Adverse events as assessed by NCI CTCAE v3.0 | All AEs will be assessed according to NCI CTCAE v3.0.
Serum alpha fetoprotein level | Serum AFP levels will be measured during the therapy, if AFP is ≥ 1.5 x ULN at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koeberle, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital - St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Koeberle D, Montemurro M, Samaras P, Majno P, Simcock M, Limacher A, Lerch S, Kovacs K, Inauen R, Hess V, Saletti P, Borner M, Roth A, Bodoky G. Continuous Sunitinib treatment in patients with advanced hepatocellular carcinoma: a Swiss Group for Clinical Cancer Research (SAKK) and Swiss Association for the Study of the Liver (SASL) multicenter phase II trial (SAKK 77/06). Oncologist. 2010;15(3):285-92. doi: 10.1634/theoncologist.2009-0316. Epub 2010 Mar 4. PMID 20203173